CLINICAL TRIAL: NCT06674187
Title: A Prospective Randomized Controlled Trial Comparing the Incidence of Parastomal Hernia After Mesenteric Molding Suturing and Non-molding Suturing in Colostomy Surgery
Brief Title: Comparing the Incidence of Parastomal Hernia After Mesenteric Molding Suturing and Non-molding Suturing in Colostomy Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yueming Sun, Dr., The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Parastomal Hernia-01
Record Dates: First submitted 2024-10-30; First posted 2024-11-05 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Parastomal Hernia
Keywords: Colostomy Surgery; Parastomal Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regular (Active Comparator): The stoma surgery will be performed using conventional non-molding suturing techniques. The specific steps include:
  1. Select an appropriate stoma site, typically within the rectus abdominis muscle.
  2. Perform routine suturing around the stoma without additional mesentery shaping.
  3. Form the stoma, ensuring a tight fit of the surrounding tissues.
  Interventions: Procedure: Mesenteric Molding Suturing Group
- Mesenteric Molding Suturing (Experimental): During the stoma surgery, the mesentery will be shaped and sutured to enhance the support around the stoma and reduce the risk of hernia formation. The specific steps include:
  1. Select an appropriate stoma site, typically within the rectus abdominis muscle.
  2. Separate the mesentery around the stoma and shape it into a sturdy support structure.
  3. Use non-absorbable sutures to fix the shaped mesentery to the abdominal wall, forming a sturdy support structure.
  4. Form the stoma on the support structure, ensuring a tight fit of the surrounding tissues.
  Interventions: Procedure: Regular

INTERVENTIONS:
Procedure: Regular — The stoma surgery will be performed using conventional non-molding suturing techniques. The specific steps include:
  1. Select an appropriate stoma site, typically within the rectus abdominis muscle.
  2. Perform routine suturing around the stoma without additional mesentery shaping.
  3. Form the stoma, ensuring a tight fit of the surrounding tissues.
  Other Names: Non-molding Suturing Group
  Arms: Mesenteric Molding Suturing
Procedure: Mesenteric Molding Suturing Group — During the stoma surgery, the mesentery will be shaped and sutured to enhance the support around the stoma and reduce the risk of hernia formation. The specific steps include:
  1. Select an appropriate stoma site, typically within the rectus abdominis muscle.
  2. Separate the mesentery around the stoma and shape it into a sturdy support structure.
  3. Use non-absorbable sutures to fix the shaped mesentery to the abdominal wall, forming a sturdy support structure.
  4. Form the stoma on the support structure, ensuring a tight fit of the surrounding tissues.
  Arms: Regular

SUMMARY:
**Research Background**

Colostomy surgery is a common surgical procedure widely used for the treatment of various gastrointestinal diseases, including rectal cancer, ulcerative colitis, and Crohn's disease. Although this surgery can significantly improve patients' quality of life and prognosis, the incidence of postoperative complications, particularly parastomal hernia (PSH), is relatively high. PSH refers to the formation of an abdominal wall hernia around the stoma, with an incidence rate that can reach up to 50%. PSH not only affects patients' quality of life but can also lead to pain, stoma dysfunction, and the need for reoperation, increasing medical costs and patient burden. Therefore, how to effectively prevent PSH has become an important topic in clinical research.

**Epidemiology of Parastomal Hernia**

The incidence of PSH varies across different studies, ranging from 10% to 50%. This variation may be due to differences in study design, patient characteristics, and surgical techniques. A systematic review and meta-analysis showed that the incidence of PSH differs significantly among different surgical techniques, with higher rates observed in traditional non-molding suturing techniques. Another large cohort study found that the incidence of PSH varies among different age groups and patients with different underlying diseases, suggesting that PSH occurrence may be influenced by multiple factors.

**Risk Factors for Parastomal Hernia**

1. **Patient Factors**:

   * **Advanced Age**: Older patients have reduced tissue elasticity and muscle strength, making them more susceptible to PSH.
   * **Obesity**: Obese patients have higher intra-abdominal pressure, increasing the risk of PSH.
   * **Smoking**: Smoking impairs wound healing, increasing the risk of PSH.
   * **Chronic Obstructive Pulmonary Disease (COPD)**: COPD patients often experience coughing and breathing difficulties, leading to increased intra-abdominal pressure and a higher risk of PSH.
   * **Diabetes**: Diabetic patients have poorer wound healing capabilities, making them more prone to PSH.
   * **Malnutrition**: Malnutrition impairs tissue repair, increasing the risk of PSH.
2. **Surgical Factors**:

   * **Surgical Technique**: Different surgical techniques have a significant impact on the incidence of PSH. Traditional non-molding suturing techniques, which lack support for the tissues around the stoma, have a higher incidence of PSH.
   * **Stoma Location**: Improper stoma placement, such as outside the rectus abdominis muscle, increases the risk of PSH.
   * **Stoma Size**: An oversized or undersized stoma can affect stoma function and increase the risk of PSH.
   * **Use of Mesh**: Using synthetic or biological mesh can significantly reduce the incidence of PSH. However, the use of mesh may bring risks of infection and other complications.
3. **Postoperative Factors**:

   * **Early Mobilization**: Appropriate early mobilization promotes circulation and wound healing, but excessive activity can increase intra-abdominal pressure and the risk of PSH.
   * **Increased Intra-abdominal Pressure**: Activities such as coughing, constipation, and heavy lifting can increase intra-abdominal pressure and the risk of PSH.
   * **Infection**: Postoperative infections can impair wound healing and increase the risk of PSH.

**Prevention Strategies for Parastomal Hernia**

1. **Improvement in Surgical Techniques**:

   * **Mesenteric Molding Suturing**: In recent years, mesenteric molding suturing has gained attention due to its potential advantages. Mesenteric molding suturing strengthens the support around the stoma, reducing the protrusion of abdominal contents and thus lowering the incidence of PSH. A retrospective study showed that patients who underwent mesenteric molding suturing had a significantly lower incidence of PSH compared to those who received traditional non-molding suturing. However, these studies are mostly retrospective and have certain biases and limitations, lacking high-quality prospective randomized controlled trials to validate these findings.
   * **Use of Mesh**: Some studies have shown that using synthetic or biological mesh can significantly reduce the incidence of PSH. The mesh provides additional support, reducing the protrusion of abdominal contents and thus lowering the risk of PSH. However, the use of mesh may bring risks of infection and other complications, requiring a careful balance of benefits and risks.
2. **Postoperative Care**:

   * **Early Mobilization Guidance**: Appropriate early mobilization promotes circulation and wound healing, but excessive activity should be avoided to prevent increased intra-abdominal pressure.
   * **Avoidance of Increased Intra-abdominal Pressure**: Patients should be advised to avoid activities that can increase intra-abdominal pressure, such as coughing, constipation, and heavy lifting.
   * **Infection Prevention**: Keeping the stoma area clean and dry and promptly managi

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patients requiring colostomy surgery.
* Ability to provide written informed consent.
* Expected survival of more than one year.
* No severe comorbidities such as heart, lung, liver, or kidney dysfunction.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* History of major abdominal surgery that could affect the development of PSH.
* Mental illness that impairs understanding of the study content and ability to give informed consent.
* Patients receiving immunosuppressive therapy or chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of PSH within one year postoperatively | 1 year
  Incidence of PSH within one year postoperatively, from CT or body check

SECONDARY OUTCOMES:
Incidence of stoma-related complications | 1 year
  stoma bleeding, stoma necrosis, and stoma prolapse through clinical observation.
Operative time and time to stoma function recovery | 1 year
  Operative time and time to stoma function recovery through questionnaire survey
Quality of life assessment | 1 year
  Quality of life assessment through questionnaire survey

IPD SHARING:
Plan to Share IPD: No